CLINICAL TRIAL: NCT01045473
Title: Prospective Study of Minimally Invasive Spinal Fusion Surgery for the Treatment of Spondylolisthesis, Degenerative Disk Disease, Spinal Stenosis and Degenerative Scoliosis
Brief Title: Prospective Study of Minimally Invasive Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Society for Minimally Invasive Spine Surgery (Other)
Responsible Party: Greg Anderson, MD, Society for Minimally Invasive Spine Surgery
Other Study IDs: SMISS-001
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Degenerative Disk Disease; Spondylolisthesis; Spinal Stenosis; Degenerative Scoliosis
Keywords: MIS; Minimally Invasive Spine Surgery; Fusion; Spine; SMISS
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The population of the US is aging. They remain more active and place greater demands on their musculoskeletal system. A key problem is that pain and disability of age related spinal disorders will increase. Problems such as Degenerative Lumbar Spondylolisthesis, Degenerative Disk Disease, Spinal Stenosis and Degenerative Scoliosis are age related problems that are treated with spinal fusion when non-operative treatment fails. Traditional open surgery poses significant risk for patients in this age group. The use of minimally invasive spinal surgery techniques provides an opportunity to treat these patients with less morbidity than traditional open surgery.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

* Patient age 21 - 90 years.
* Diagnosis of Spondylolisthesis, degenerative disk disease, and degenerative scoliosis (any curve magnitude).
* A spinal fusion is being undertaken via the minimally invasive approach.
* The patient agrees to follow-up for routine care for at least 2 years post-operatively.

Exclusion Criteria:

* Inability for post-operative follow-up

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthropedic surgeon's clinic. Neurosurgeon's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

REFERENCES:
- See also: Related Info — http://www.smiss.org